CLINICAL TRIAL: NCT01014117
Title: A Phase I Study to Evaluate Single and Multiple (Seven) Oral Doses of SRT2104 on the Endotoxin Induced Inflammatory Response in Healthy Male Subjects
Brief Title: Effect of SRT2104 on Endotoxin-induced Inflammation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 114009
Record Dates: First submitted 2009-11-12; First posted 2009-11-16 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — SRT2104

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): The Placebo treatment group will be administered eight oral placebo capsules once daily for 7 days.
  A trained investigative site member will administer the test material to subjects on Day 1, 2, and 7. On Days 1, 2 and 7 the subjects will receive SRT2104 or placebo approximately 15min following the consumption of a standardized meal at the study center. During non-clinic days, the subject will self-administer the test material approximately 15 min following consumption of a standardized meal at home. Test material should be administered with approximately 400mL of water. On Days 1 and 7, dosing will occur at approximately 7AM. Dosing on Days 2-6 will occur before 9AM. Subjects must wait at least 1-2 hrs after dosing before consuming additional calories on all dosing days.
  Interventions: Drug: Placebo
- Placebo and 2.0g SRT2104 (Active Comparator): This treatment group will be administered eight oral placebo capsules once daily for 6 days followed by 2.0g SRT2104 administered as eight oral SRT2104 capsules on Day 7. A trained investigative site member will administer the test material to subjects on Day 1, 2, and 7. On Days 1, 2 and 7 the subjects will receive SRT2104 or placebo approximately 15min following the consumption of a standardized meal at the study center. During non-clinic days, the subject will self-administer the test material approximately 15 min following consumption of a standardized meal at home. Test material should be administered with approximately 400mL of water. On Days 1 and 7, dosing will occur at approximately 7AM. Dosing on Days 2-6 will occur before 9AM. Subjects must wait at least 1-2 hrs after dosing before consuming additional calories on all dosing days.
  Interventions: Drug: Placebo; Drug: SRT2104
- 2.0g SRT2104 (Active Comparator): The 2.0g SRT2104 treatment group will be administered eight oral SRT2104 capsules once daily for 7 days. A trained investigative site member will administer the test material to subjects on Day 1, 2, and 7. On Days 1, 2 and 7 the subjects will receive SRT2104 or placebo approximately 15min following the consumption of a standardized meal at the study center. During non-clinic days, the subject will self-administer the test material approximately 15 min following consumption of a standardized meal at home. Test material should be administered with approximately 400mL of water. On Days 1 and 7, dosing will occur at approximately 7AM. Dosing on Days 2-6 will occur before 9AM. Subjects must wait at least 1-2 hrs after dosing before consuming additional calories on all dosing days.
  Interventions: Drug: SRT2104

INTERVENTIONS:
Drug: Placebo — Matching placebo will be supplied as hard gelatin capsules, with each containing an appropriate amount of placebo.
  Arms: Placebo; Placebo and 2.0g SRT2104
Drug: SRT2104 — SRT2104 will be supplied as hard gelatin capsules, with each containing 250mg of SRT2104.
  Arms: 2.0g SRT2104; Placebo and 2.0g SRT2104

SUMMARY:
SRT2104 is a potent small molecule activator of SIRT1 that has been found to inhibit systemic inflammation induced by intravenous injection of lipopolysaccharide (LPS) in mice. The objective of this study is to test if SRT2104 may be a novel compound for the treatment of inflammatory disorders in man.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination and laboratory tests carried out within 28 days prior to day 1. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures
* Male between 18 and 35 years of age inclusive, at the time of signing the informed consent
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* No history of HIV 1 and 2, and hepatitis B and C
* Normal 12 lead ECG without any clinically significant abnormality as judged by the Investigator and average QTcB or QTcF < 450 msec
* Normal renal and liver function (normal serum creatinine and liver function tests (ALT, AST, Total bilirubin, alkaline phosphatase)
* Subjects must agree with their partners to use double-barrier birth control or abstinence while participating in the study and for 12 weeks following the last dose of study drug

Exclusion Criteria:

* As a result of the medical interview, physical examination or screening investigations, the Investigator or appropriately qualified designee considers the subject unfit for the study
* Subject has had a major illness in the past three months or any significant chronic medial illness that the investigator would deem unfavourable for enrolment including inflammatory diseases
* Subjects with a history of any type of malignancy with the exception of successfully treated basal cell cancer of the skin
* Subject has renal impairment
* Subject has a past or current gastro-intestinal disease which may influence drug absorption
* The subject has a known positive test for hepatitis C antibody or hepatitis B surface antigen
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* The subject has a known positive test for HIV antibody 1 or 2
* Subject has a history, within three years, of drug abuse (including benzodiazepines, opioids, amphetamine, cocaine, THC) or a positive drug results at the Screening visit
* History of alcoholism and/or is drinking more than 3 drinks per day. Alcoholism is defined as an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits
* The subject has participated in a clinical trial and has received an investigational product within three months of the first dosing day in the current study
* Use of prescription or non-prescription drugs, and herbal and dietary supplements within 7 days unless in the opinion of the Investigator and Medical Monitor the medication will not interfere with the study procedures or compromise subject safety
* Subject has difficultly in donating blood or accessibility of a vein in left or right arm
* Subject has donated more than 350 mL of blood in last 3 months
* Subject uses tobacco products
* Any other issue that, in the opinion of the Principal Investigator, would could be harmful to the subject or compromise interpretation of the data

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2009-12-09 (Actual); Primary Completion 2010-05-10 (Actual); Study Completion 2010-05-10 (Actual)

PRIMARY OUTCOMES:
To determine if a single or 7 daily doses of SRT2104 attenuates the inflammatory response in normal healthy male subjects after exposure to low-dose endotoxin (LPS). | Measurements of inflammation will be conducted on plasma samples obtained on Day7 at -3, 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12hrs. Samples will also be taken on Day8, approximately 24hrs after dosing on Day7.

SECONDARY OUTCOMES:
To determine PK of SRT2104 in normal healthy male subjects exposed to low-dose endotoxin (LPS). | Plasma samples will be collected at pre-dose, 15min, 30min, and 1, 2, 3, 4, 8, and 12hrs post-dose on Day1 and Day7. Plasma samples will also be collected on Day2 and Day8 and at 24hrs post-dose Day1 and Day7, respectively.
To determine the safety profile of SRT2104 in healthy male subjects exposed to low-dose endotoxin (LPS). | Safety will be monitored by AEs, VS, physical exam, labs and ECGs during the course of the study.
To determine the effect of SRT2104 on other parameters following low-dose endotoxin (LPS) exposure in humans e.g., lipid profile, serum amyloid phospholipids, metabolic profiles and gene expression analysis etc. | Blood samples will be collected for exploratory gene expression analysis pre-dose on Days1 and 7, and 4hrs after LPS exposure on Day7. Samples for other parameters will be collected during fasting, pre-dose on Days1 and 7 and 24hrs post-dose on Day8.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] van der meer, AJ, Scicluno, B, Lin, J, Jacobson, EW, Vlasuk, GP, van der Poll. The first demonstration of clinical activity by a small molcule SIRT1 activator: SRT 2104 reduces cytokine release and coagulation activation in a human enotoxin model. [Inflammation Research]. 2011;60(Supplement 1):S1-321.
- [Derived] van der Meer AJ, Scicluna BP, Moerland PD, Lin J, Jacobson EW, Vlasuk GP, van der Poll T. The Selective Sirtuin 1 Activator SRT2104 Reduces Endotoxin-Induced Cytokine Release and Coagulation Activation in Humans. Crit Care Med. 2015 Jun;43(6):e199-202. doi: 10.1097/CCM.0000000000000949. PMID 25978169
- See also: Results for study 114009 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114009?search=study&study_ids=114009#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 114009 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114009 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114009 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114009 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114009 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114009 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register